CLINICAL TRIAL: NCT02517463
Title: Observational Study on the Clinical Efficacy of Ulipristal for Emergency Contraception When Administered Before or After Ovulation
Brief Title: Ulipristal Emergency Contraception Used Before or After Ovulation
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Collaborators: The Family Planning Association of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Hang Wun Raymond Li, Clinical Associate Professor, The University of Hong Kong
Other Study IDs: UW10-392
Record Dates: First submitted 2015-08-03; First posted 2015-08-07 (Estimated); Results first posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2017-10

CONDITIONS: Contraception
Keywords: Emergency contraception; ulipristal acetate; efficacy
MeSH Terms: interventions — ulipristal acetate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pre-ovulatory: Ulipristal acetate 30 mg single oral dose
  Interventions: Drug: Ulipristal acetate
- Post-ovulatory: Ulipristal acetate 30 mg single oral dose
  Interventions: Drug: Ulipristal acetate

INTERVENTIONS:
Drug: Ulipristal acetate — This is an observational study on subjects taking a single intervention, i.e. ulipristal acetate for emergency contraception. The intervention is not randomised nor assigned by the investigator.
  Other Names: Ella

SUMMARY:
This was a prospective, open-label, single-drug, uncontrolled, observational clinical study.

Women attending the Family Planning Association of Hong Kong (FPAHK) for emergency contraception within 120 hours of UPSI were recruited. Subjects were recruited from both the Birth Control Clinics and Youth Health Care Centres of the FPAHK.

Depending on the timing in relation to ovulation in the current menstrual cycle at the time of presentation, the women were classified into two groups:

Group 1: pre-ovulatory Group 2: post-ovulatory

After counseling and obtaining informed consent, eligible subjects received a single dose of ulipristal acetate 30 mg (ellaOne®) under direct supervision. A baseline blood test for hormonal profile (LH, oestradiol and progesterone) and ultrasound scan for ovarian follicle assessment were carried out by a designated doctor or research nurse at the clinic visit.

The subjects were advised not to have further acts of coitus before the return of menstruation. They were given a diary chart to record vaginal spotting and bleeding, possible side effects and further acts of intercourse, if any, and the contraceptive method used. A follow-up appointment were be arranged about 1-2 weeks after the expected next menstruation. Any events of unplanned pregnancy and adverse effects were recorded for analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy women aged 18 years or above;
2. Regular menstrual cycles (every 21-35 days) within the past three cycles;
3. Requesting emergency contraception within 120 h of a single act of unprotected intercourse in the current menstrual cycle;
4. Willing to abstain from further acts of unprotected intercourse and;
5. Available for follow-up over the next 6 weeks

Exclusion Criteria:

1. Post-abortion or postpartum patients whose period had not yet returned
2. Regular use of prescription drugs before admission to the study and
3. Intercourse during the treatment cycle more than 120 h before admission into the study.
4. Found pregnant at the time of presentation
5. Breastfeeding women
6. Women who have been sterilized (or partner being sterilized) or have intrauterine contraceptive device in-situ
7. Uncertain about the date of the last menstrual period
8. Women who had used hormonal contraceptive in the current or past one cycle

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 700 women attending the Family Planning Association of Hong Kong for emergency contraception who fulfilled the inclusion criteria and not meeting the exclusion criteria were recruited.
Sampling Method: Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2011-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hang Wun Raymond Li, MBBS, FRCOG, Principal Investigator — The University of Hong Kong

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 700 women were recruited at a community family planning clinic of the Family Plannng Association of Hong Kong, Hong Kong, between May 2011 and March 2014
Period: Overall Study
Arm/Group | Pre-ovulatory | Post-ovulatory
Started | 369 | 331
Completed | 364 | 329
Not Completed | 5 | 2
Not completed — Lost to Follow-up | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-ovulatory | Post-ovulatory | Total
Number analyzed (Participants) | 364 | 329 | 693
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 364 | 329 | 693
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 31 [28 to 37] | 34 [28 to 39] | 32 [28 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 364 | 329 | 693
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 355 | 322 | 677
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 7 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Hong Kong | 364 | 329 | 693

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Pregnancies Prevented (PPP)
Time Frame: one cycle (i.e. up to about 4 weeks)
Measure: Number; unit: percentage of pregnancies prevented
Arm/Group | Pre-ovulatory | Post-ovulatory
Number analyzed (Participants) | 364 | 329
percentage of pregnancies prevented | 77.5 | 36.9
Statistical Analysis 1: Comparison: Pre-ovulatory vs Post-ovulatory; Test type: Non-Inferiority or Equivalence — The PPP from a previous study was 67.2%. Assuming the PPP in the "preovulatory" and "post-ovulatory" groups were equivalent, and taking 10% to be the maximum permitted difference for equivalence, a minimum of 273 subjects in each group would be required to confirm equivalence between the two groups with a power of 80% and type I error of 0.05. Therefore, our recruitment of 700 subjects with more than 300 in each group was sufficient; p < 0.0001, Chi-squared

2. Secondary Outcome: Failure Rate
Description: Number of subjects who got pregnant / Total number of subjects in the group
Time Frame: one cycle (i.e. up to about 4 weeks)
Measure: Number; unit: percentage of participants
Arm/Group | Pre-ovulatory | Post-ovulatory
Number analyzed (Participants) | 364 | 329
percentage of participants | 1.4 | 2.1
Statistical Analysis 1: Comparison: Pre-ovulatory vs Post-ovulatory; Test type: Superiority or Other; p = 0.564, Fisher Exact

3. Secondary Outcome: Change in the Length of the Index Menstrual Cycle From Baseline
Description: shortening or lengthening of the index menstrual cycle compared to the previous menstrual pattern of the subject
Time Frame: one cycle (i.e. up to about 4 weeks)
Population: Only subjects with follow-up information were included in this part of analysis
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Pre-ovulatory | Post-ovulatory
Number analyzed (Participants) | 355 | 322
days | 3 [0 to 6] | -1 [-3 to 1]
Statistical Analysis 1: Comparison: Pre-ovulatory vs Post-ovulatory; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Pre-ovulatory | Post-ovulatory
Serious Adverse Events (participants affected / at risk) | 0/364 | 0/329
Other Adverse Events (participants affected / at risk) | 117/364 | 111/329
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-ovulatory (N=364) | Post-ovulatory (N=329)
Minor complaints (General disorders) | 117 | 111

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No